CLINICAL TRIAL: NCT01450072
Title: Prospective Randomized Endovascular Therapy in Multiple Sclerosis - PREMiSE
Acronym: PREMiSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Adnan H. Siddiqui, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSG1730210B
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Sham Comparator): Venography and sham angioplasty
  Interventions: Other: Control arm
- Active arm (Active Comparator): therapeutic balloon angioplasty
  Interventions: Device: Selective Venography followed by therapeutic balloon angioplasty

INTERVENTIONS:
Device: Selective Venography followed by therapeutic balloon angioplasty — Venography followed by therapeutic balloon angioplasty
  Arms: Active arm
Other: Control arm — Venography and sham angioplasty
  Arms: Control arm

SUMMARY:
The Departments of Neurology and Neurosurgery are conducting this research study to evaluate the safety and effectiveness of intravascular angioplasty for the treatment of venous narrowing in the treatment of Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* EDSS 0-6.5 (0-5.5 in the phase II of the study)
* Diagnosis of relapsing MS according to the McDonald criteria (Polman et al., 2005)
* 1 relapse within the past 12 months or GAD positive lesion on an MRI within the past 3 months (only for phase II of the study)
* Be on treatment with currently FDA approved disease-modifying treatments (excluding Tysabri or steroids (within the last 30 days prior to enrollment)
* Evidence of ≥2 sonographic parameters of suspicious abnormal extracranial cerebral venous outflow (see Table 1 background and 1.5 section)
* Normal renal function: creatinine clearance level of >60

Exclusion Criteria:

* Relapse, disease progression and Tysabri and steroid treatment in the 30 days preceding study entry
* Pre-existing medical conditions known to be associated with brain pathology (e.g., neurodegenerative disorder, cerebrovascular disease, positive history of alcohol abuse, etc.)
* Severe peripheral chronic venous insufficiency
* Abnormal renal function
* Contrast allergy (anaphylaxis)
* Not accepting to undergo the endovascular treatment
* Peripheral Vascular Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Siddiqui, MD, PhD, Principal Investigator — University at Buffalo Neurosurgery
Locations (1):
- University at Buffalo Neurosurgery, Buffalo, New York, United States

REFERENCES:
- [Derived] Siddiqui AH, Zivadinov R, Benedict RH, Karmon Y, Yu J, Hartney ML, Marr KL, Valnarov V, Kennedy CL, Ramanathan M, Ramasamy DP, Dolic K, Hojnacki DW, Carl E, Levy EI, Hopkins LN, Weinstock-Guttman B. Prospective randomized trial of venous angioplasty in MS (PREMiSe). Neurology. 2014 Jul 29;83(5):441-9. doi: 10.1212/WNL.0000000000000638. Epub 2014 Jun 27. PMID 24975855

RESULTS

PARTICIPANT FLOW:
Groups:
- Venography & Sham Angioplasty: Venography and sham angioplasty
  Control arm: Venography and sham angioplasty
- Therapeutic Balloon Angioplasty: therapeutic balloon angioplasty
  Selective Venography followed by therapeutic balloon angioplasty: Venography followed by therapeutic balloon angioplasty
Period: Overall Study
Arm/Group | Venography & Sham Angioplasty | Therapeutic Balloon Angioplasty
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Active Arm | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (10.5) | 43.3 (8.2) | 44.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Immediate and Short-term SAE
Description: Percent (%) of patients with Severe Adverse Events (SAE) measured at 1 month (Short term) post-surgical safety outcome in MS patients diagnosed with CCSVI that underwent therapeutic angioplasty. The 95% confidence interval of the SAE rates for immediate and short terms will be obtained by the exact method, respectively. The immediate and short term SAE rates will be analyzed, respectively, using the Fisher's exact test.
Time Frame: 24 hours-1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Active Arm
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With More Than 75% of Normal Outflow at 1 Year Post-angioplasty
Description: Restoration of venous outflow (more than 75% of normal outflow) as measured by the combined ECD/TCD and MRV at 1 year following the angioplasty as compared to baseline as well as compared to a parallel control group of MS patients that will undergo only selective venography without balloon angioplasty (sham-angioplasty). These comparisons will be accomplished by the hierarchical linear model which takes into account the correlation within subjects. Based on the residuals, we will check the normality assumptions by the normal quantile plot and skewness.
Time Frame: 1 month, 3 months, 6 months, and 1 year post-angioplasty
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Active Arm
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Arm | Active Arm
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/10 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=10) | Active Arm (N=9)
Immune thrombocytopenic purpura (Immune system disorders) | 1 (1) | 0 (0) — Immune thrombocytopenic purpura treated with 100mg prednisone once daily
Bladder infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Bladder infection treated with antibiotics over 10 days
Shingles (Nervous system disorders) | 1 (1) | 0 (0) — Diagnosis of shingles treated with Valtrex (GlaxoSmithKline) 3x daily for 7 days
Cardiac event (Cardiac disorders) | 0 (0) | 1 (1) — Cardiac event treated with pacemaker installation
Swelling & Soreness (General disorders) | 0 (0) | 1 (1) — Swelling and soreness at left side of the neck; no treatment required
Transobturator sling (Renal and urinary disorders) | 0 (0) | 1 (1) — Hospitalization for scheduled transobturator sling procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No